CLINICAL TRIAL: NCT02309255
Title: The NOR-COR (NORwegian CORonary) Study: Identification of CHD Patients With Poor Adherence to Secondary Prevention and Their Perceived Needs for Follow-up
Brief Title: The NOR-COR Study for Coronary Prevention
Status: Completed | Type: Observational
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: The Hospital of Vestfold (Other); Oslo University Hospital (Other); Kalmar County Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NOR-COR REK ID 2013/1885
Record Dates: First submitted 2014-11-24; First posted 2014-12-05 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Secondary Coronary Prevention
Keywords: Secondary coronary prevention; Psychosocial factors; Cardiac rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Salvia for genetic analyses
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- coronary heart disease patients
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
The NOR-COR study is a cross-sectional, observational study designed to explore a large number of cardiovascular, inflammatory, genetic, behavioral, and psychosocial factors (including anxiety, depression, quality of life) in 1369 patients with established coronary heart disease (CHD) hospitalized in the Sections for Cardiology at the hospitals in Drammen (n=722) and Vestfold (n=647). Study data from an extensive questionnaire, clinical and laboratory data, and sputum/saliva for genetic analyses will be collected.

The main overall aim of the NOR-COR study is to develop new strategies to improve secondary prevention for underserved high risk patient-groups with CHD. The first study phase aims to collect information necessary to develop empirically based future secondary coronary prevention interventions. In a genetic sub-project markers associated with CHD and personality type will be explored.

The study will evaluate current secondary preventive programs and explore the mechanisms that link behavioral, psychosocial, inflammatory, and genetic factors to poor prognosis. The study will in short term provide new knowledge potentially useful for increasing participation in current cardiac rehabilitation/secondary preventive programs. For a longer perspective these associations may be useful for design of new intervention programs to selected high risk patient groups whom may be in need of programs with different content and/or of longer duration than those currently being applied.

ELIGIBILITY:
Inclusion criteria:

All patients aged 18-80 years with first or recurrent diagnosis or treatments for CHD: a) acute myocardial infarction [ICD-10; I21], b) coronary artery by-pass graft operation (CABG), or c) elective or emergency PCI [ICD-10; I25]) have been identified from hospital patient discharge lists (diagnostic lists) by searching chronologically after last admission the past three years. In patients with recurrent diagnosis the last event will define the event.

Exclusion Criteria:

* Cognitive impairment that would invalidate assessment including all patients living at nursing home and psychosis.
* Short life expectancy (i.e. <1 year) due to terminal heart (NYHA class 4), lung (chronic obstructive pulmonary disease GOLD 4)-, liver- or kidney disease (chronic kidney disease stage 5), malignant disease, or other reason.
* Not able to understand and write the Norwegian language or refuse to give written informed consent to study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1365 CHD patients
Sampling Method: Probability Sample
Enrollment: 975 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Cardiovascular risk factors, lifestyle, and drug adherence | Within 2 years after study inclusion

SECONDARY OUTCOMES:
Readmission with a coronary event, acute myocardial infarctrion and cardiovascular mortality | Within 5 years after study inclusion

OTHER OUTCOMES:
The hospital anxiety and depression scale (HADS) | Within 2 years after study inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Vestre Viken HF, Drammen Hospital and The Hospital of Vestfold, Drammen and Tønsberg, Buskerud and Vestfold, Norway

REFERENCES:
- [Derived] Sverre E, Peersen K, Perk J, Husebye E, Gullestad L, Dammen T, Otterstad JE, Munkhaugen J. Challenges in coronary heart disease prevention - experiences from a long-term follow-up study in Norway. Scand Cardiovasc J. 2021 Apr;55(2):73-81. doi: 10.1080/14017431.2020.1852308. Epub 2020 Dec 4. PMID 33274648
- [Derived] Sverre E, Peersen K, Weedon-Fekjaer H, Perk J, Gjertsen E, Husebye E, Gullestad L, Dammen T, Otterstad JE, Munkhaugen J. Preventable clinical and psychosocial factors predicted two out of three recurrent cardiovascular events in a coronary population. BMC Cardiovasc Disord. 2020 Feb 5;20(1):61. doi: 10.1186/s12872-020-01368-6. PMID 32024471
- [Derived] Munkhaugen J, Hjelmesaeth J, Otterstad JE, Helseth R, Sollid ST, Gjertsen E, Gullestad L, Perk J, Moum T, Husebye E, Dammen T. Managing patients with prediabetes and type 2 diabetes after coronary events: individual tailoring needed - a cross-sectional study. BMC Cardiovasc Disord. 2018 Aug 3;18(1):160. doi: 10.1186/s12872-018-0896-z. PMID 30075751
- [Derived] Sverre E, Otterstad JE, Gjertsen E, Gullestad L, Husebye E, Dammen T, Moum T, Munkhaugen J. Medical and sociodemographic factors predict persistent smoking after coronary events. BMC Cardiovasc Disord. 2017 Sep 6;17(1):241. doi: 10.1186/s12872-017-0676-1. PMID 28877684
- [Derived] Sverre E, Peersen K, Husebye E, Gjertsen E, Gullestad L, Moum T, Otterstad JE, Dammen T, Munkhaugen J. Unfavourable risk factor control after coronary events in routine clinical practice. BMC Cardiovasc Disord. 2017 Jan 21;17(1):40. doi: 10.1186/s12872-016-0387-z. PMID 28109259